CLINICAL TRIAL: NCT00771901
Title: Effect of Endoplasmic Reticulum Stress on Metabolic Function
Acronym: TUDCA/PBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 07-1114
Record Dates: First submitted 2008-10-10; First posted 2008-10-15 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-04

CONDITIONS: Insulin Resistance; Diabetes; Obesity
Keywords: obesity; insulin resistance; type II diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus; Obesity; Diabetes Mellitus, Type 2 | interventions — ursodoxicoltaurine; 4-phenylbutyric acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects will be given a placebo rather than tauroursodeoxycholic acid.
  Interventions: Other: placebo
- tauroursodeoxycholic acid (Experimental): Subjects will receive tauroursodeoxycholic acid for four weeks.
  Interventions: Drug: tauroursodeoxycholic acid
- PBA (Experimental): Subjects will receive sodium phenylbutyrate for four weeks.
  Interventions: Drug: sodium phenylbutyrate

INTERVENTIONS:
Drug: tauroursodeoxycholic acid — 1750 mg/day for four weeks. Seven pills daily, 2 with breakfast, 2 with lunch, and 3 with dinner.
  Other Names: TUDCA
  Arms: tauroursodeoxycholic acid
Other: placebo — 7 pills daily for 4 weeks
  Arms: Placebo
Drug: sodium phenylbutyrate — 20g/day for four weeks.
  Other Names: PBA
  Arms: PBA

SUMMARY:
Normally, the hormone insulin works to help keep blood sugar normal. However, as a person gains weight, insulin does not work as well and blood sugar tends to be a little higher than normal. This is called "insulin resistance".

Two investigational drugs (not approved by the Food and Drug Administration) for the treatment of high lipid levels or insulin resistance are being examined in this study: one drug is called tauroursodeoxycholic acid (TUDCA), the other is called sodium phenylbutyrate (PBA). This study is designed to test if TUDCA and/or PBA is effective in people who are obese with insulin resistance and high lipids. We hypothesize that pharmacologically-induced decreases in ER stress will improve insulin action and hepatic lipid metabolism in obese subjects.

DETAILED DESCRIPTION:
A 4-week randomized, controlled trial will be conducted to evaluate the following specific aims in obese subjects:

Determine the effect of treatment with TUDCA or PBA on:

1. Body fat distribution: a) intrahepatic triglyceride (IHTG) content, b) intramyocellular triglyceride (IMTG) content, and c) intra-abdominal fat content, assessed by using magnetic resonance spectroscopy and magnetic resonance imaging.
2. In vivo insulin sensitivity in adipose tissue (suppression of lipolysis), liver (suppression of glucose production), and skeletal muscle (stimulation of glucose uptake), assessed by using the hyperinsulinemic-euglycemic clamp procedure in conjunction with stable isotope tracer infusion.
3. VLDL-triglyceride (TG) and VLDL-apolipoprotein-B100 (apoB-100) secretion rates, assessed by stable isotopically labeled tracer infusion methods.
4. Skeletal muscle intracellular insulin signaling, fatty acid oxidation, and markers of inflammation, assessed by evaluating skeletal muscle biopsies ex vivo.
5. Adipose tissue insulin signaling, ER stress, and inflammation, assessed by evaluating adipose tissue biopsies ex vivo.

ELIGIBILITY:
Inclusion Criteria:

* BMI range 30 to 45
* sedentary (defined as regular exercise < 1 h per week or < 2 x/week for the last 6 months)

Exclusion Criteria:

* active or previous infection with hepatitis B or C
* liver diseases
* history of alcohol abuse
* current alcohol consumption > 20 g/day
* severe hypertriglyceridemia ( > 400 mg/dL)
* active peptic ulcer disease
* taking cholestyramine or oral contraceptives
* women who are pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Kars M, Yang L, Gregor MF, Mohammed BS, Pietka TA, Finck BN, Patterson BW, Horton JD, Mittendorfer B, Hotamisligil GS, Klein S. Tauroursodeoxycholic Acid may improve liver and muscle but not adipose tissue insulin sensitivity in obese men and women. Diabetes. 2010 Aug;59(8):1899-905. doi: 10.2337/db10-0308. Epub 2010 Jun 3. PMID 20522594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants will be recruited by reviewing the VFH database pf research subjects and by local postings. Potential subjects will be contacted by telephone for an initial pre-screen, at which time the study is discussed and a brief medical history and concomitant medication list is obtained. ICF will be sent to interested subjects.
Pre-assignment Details: Screening tests to determine eligibility included: medical hx & PE, blood tests, resting ECG, OGTT, MRI/MRS/MRE of abdomen/liver, and DEXA scan. Two baseline metabolism studies prior to study drug intervention. There were 67 screen fails, 4 subjects withdrew consent before beginning study intervention.
Groups:
- Sodium Phenylbutyrate: Subjects will receive sodium phenylbutyrate for four weeks.
  sodium phenylbutyrate: 20g/day for four weeks.
Period: Overall Study
Arm/Group | Placebo | Tauroursodeoxycholic Acid | Sodium Phenylbutyrate
Started | 10 | 10 | 10
Completed | 10 | 10 | 6
Not Completed | 0 | 0 | 4
Not completed — Dissat w/# of study medication (40/day) | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tauroursodeoxycholic Acid | Sodium Phenylbutyrate | Total
Number analyzed (Participants) | 10 | 10 | 6 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 6 | 26
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (14) | 47 (9) | 49 (8) | 47 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 2 | 14
  Male | 4 | 4 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Body Composition
Description: Fat mass (%)
Time Frame: Baseline and four weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Placebo | Tauroursodeoxycholic Acid | Sodium Phenylbutyrate
Number analyzed (Participants) | 10 | 10 | 6
percentage
  Before Intervention | 39 (7) | 39 (8) | 37 (6)
  After Intervention | 39 (7) | 39 (8) | 39 (7)

2. Secondary Outcome: Insulin Sensitivity in the Liver
Description: HISI (hepatic insulin sensitivity index). HISI is the inverse of the product of endogenous glucose production and plasma insulin concentration and provides an index of how well circulating insulin controls the amount of glucose supplied by the liver. A higher number is indicative of greater insulin sensitivity.
Time Frame: Baseline and four weeks
Measure: Mean (Standard Deviation); unit: 100/ (µmol/min * uIU/mL)
Arm/Group | Placebo | Tauroursodeoxycholic Acid | Sodium Phenylbutyrate
Number analyzed (Participants) | 10 | 10 | 7
100/ (µmol/min * uIU/mL)
  Before Intervention | 0.010 (0.007) | 0.009 (0.004) | 0.008 (0.003)
  After Intervention | 0.008 (0.004) | 0.012 (0.006) | 0.009 (0.003)

3. Secondary Outcome: VLDL-triglyceride (TG) Concentration
Time Frame: Baseline and four weeks
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Placebo | Tauroursodeoxycholic Acid | Sodium Phenylbutyrate
Number analyzed (Participants) | 7 | 8 | 5
mmol/l
  Before Intervention | 0.57 (0.33) | 0.74 (0.50) | 0.89 (0.25)
  After Intervention | 0.58 (0.33) | 0.75 (0.56) | 0.97 (0.18)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time participants signed the informed consent until 30 days after study completion.
Arm/Group | Placebo | Tauroursodeoxycholic Acid | Sodium Phenylbutyrate
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes